CLINICAL TRIAL: NCT02936843
Title: Targeting Inflammation With Salsalate in Type 1 Diabetes Neuropathy-TINSAL -T1DN
Brief Title: Targeting Inflammation With Salsalate in Type 1 Diabetes Neuropathy
Acronym: TINSAL-T1DN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Rodica Pop-Busui, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00103828
Record Dates: First submitted 2016-06-30; First posted 2016-10-18 (Estimated); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes; Peripheral Neuropathy
Keywords: Pain; Inflammation; Diabetes Mellitus; Adult; Neuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Peripheral Nervous System Diseases; Pain; Inflammation; Diabetes Mellitus | interventions — salicylsalicylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Salsalate (Experimental): Salsalate, 1 gram by mouth, 3 times daily (3 grams per day) for 12 months.
  Interventions: Drug: Salsalate
- Comparator (Placebo Comparator): Placebo for Salsalate, 2 tablets by mouth, 3 times daily for 12 months
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Salsalate — 1 gram, 3 times daily by mouth (total of 3 grams daily)
  Other Names: disalcid
  Arms: Salsalate
Drug: PLACEBO — Placebo for Salsalate; 2 Tablets, 3 times daily by mouth (total of 3 grams daily)
  Arms: Comparator

SUMMARY:
Diabetic neuropathy (DN) is the most common chronic complication of diabetes, affecting up to50% of individuals with type 1 diabetes (T1DM).

Multiple pre-clinical and clinical studies demonstrate a pathogenic role for inflammation, especially cytokine production, in the disease course of DN and CAN. This suggests that agents with known anti-inflammatory properties, such as salicylates, may prevent the development of DN and the pain associated with DN. This study builds upon and expands on prior work done by the investigators with salsalate, a pro-drug form of salicylate, as an agent to address inflammatory pathways in people with T1DM.

DETAILED DESCRIPTION:
Diabetic neuropathy (DN) is the most common chronic complication of diabetes, affecting up to50% of individuals with type 1 diabetes (T1DM). DN is a progressive disease, leading to severe morbidity and staggering health care costs. Patients experience poor quality of life due to pain, loss of sensation leading to poor balance, falls and eventual foot deformities with high rates of ulcerations and amputations. While not as commonly diagnosed as DN, cardiovascular autonomic neuropathy (CAN) carries equal morbidity with patients experiencing orthostasis, arrhythmias and premature death).

Despite the high morbidity associated with DN, most randomized clinical trials evaluating therapies for established DN have been disappointing. To date there is no pathogenetic treatment for this condition. The Diabetes Control and Complications Trial (DCCT) demonstrated that intensive control designed to achieve near-normal glycemia is essential in reducing the risk of DN development in type 1 diabetes (8, 9). However, attainable intensive glycemic control, although necessary, is insufficient to prevent adverse nervous system effects, justifying a therapeutic need to identify new drug targets to treat DN early in its course. One such new therapeutic target is inflammation. Multiple pre-clinical and clinical studies demonstrate a pathogenic role for inflammation, especially cytokine production, in the disease course of DN and CAN. This suggests that agents with known anti-inflammatory properties, such as salicylates, may prevent the development of DN and the pain associated with DN. Salsalate, a pro-drug form of salicylate, is a FDA approved drug commonly indicated for relief of the signs and symptoms of rheumatoid arthritis, osteoarthritis and related rheumatic disorders. In vitro and in vivo studies and human trials have shown that salicylate therapy is effective in controlling low grade inflammation in diabetes by inhibition of the inhibitor of the κB kinase (IKKβ)/NF-κB pathway. It has a large margin of safety (unlike other salicylates), and a low cost. There is also extensive experience with long-term human use of salsalate.

Several studies show that salsalate causes no greater intestinal occult blood loss than placebo and has no suppressive effects on renal prostaglandin production in contrast to aspirin or NSAIDs. The recently published NIDDK-funded "Targeting Inflammation Using Salsalate in Type 2 Diabetes (TINSAL-T2D)" trial confirmed salutary effects of 3.5 gram/day salsalate on markers of inflammation, glucose control and overall safety after 48 weeks patients with type 2 diabetes. The Investigators' initial NIDDK funded R03 (DK 094499) grant confirmed the safety and feasibility of targeting inflammation with salsalate treatment in T1DM subjects with DN. The Investigators' current study builds upon and expands their initial promising results and will either confirm or refute the therapeutic efficacy of salsalate in a larger T1DM cohort.

ELIGIBILITY:
Inclusion Criteria

1. T1DM;
2. age 18-70;
3. mild DN as defined by symptoms and/or signs, confirmed by at least one abnormality in electrophysiology studies (abnormality of at least one attribute among conduction velocity, latency, amplitude or F-Wave in at least one nerve among sural sensory, ulnar sensory, or peroneal motor);
4. sural nerve amplitude > 0 μV. If sural nerve amplitude is 0 μV (unrecordable) peroneal motor nerve conduction velocity must be ≥ 35 m/second*;
5. on a stable insulin regimen for the 3 months prior to enrollment;
6. be willing and capable of signing the IRB approved consent form and willing and able to cooperate with the medical procedures for the study duration;
7. be willing to accept random treatment assignment to salsalate or placebo; and
8. women of childbearing age agree to use an appropriate contraceptive method (hormonal, IUD, or diaphragm) for the duration of the study and must have a negative urine pregnancy test at screening.

Exclusion Criteria

1. history of severe DN, active lower limb ulceration or lower limb amputation directly caused by diabetic neuropathy, or risk factors for any other causes of neuropathy (e.g. active hepatitis C, end stage renal disease, systemic lupus erythematosus or a known hereditary neuropathy) as determined through medical history, family history, history of medications, occupational history, history of exposure to toxins, physical and neurological examinations);
2. history of recent severe hypoglycemia (within prior 6 months) as defined by hypoglycemia resulting in coma or seizure or a history of recurrent diabetic ketoacidosis (DKA) or any diabetic ketoacidosis within the last three months.
3. history of persistent macroalbuminuria [random urine microalbumin creatinine ratio (ACR) >300 mg/gm]. ACR up to 300 mg/gm is acceptable if serum creatinine is <1.4 for women, <1.5 for men AND estimated GFR (eGFR) is > 60;
4. serum creatinine >1.4 for women and >1.5 for men or eGFR <60 [possible chronic kidney disease stage 3 or greater calculated using the Modification of Diet in Renal Disease (MDRD) equation];
5. pregnancy or lactation, or intention to become pregnant in next 12 months;
6. history of previous lung, kidney, pancreas, liver, cardiac or bone marrow transplant;
7. history of drug or alcohol abuse within the previous 5 years, or current weekly alcohol consumption >10 units/week;
8. use of warfarin (Coumadin), clopidogrel (Plavix), dipyridamole (Persantine), heparin or other anticoagulants, probenecid (Benemid, Probalan), sulfinpyrazone (Anturane) or other uricosuric agents; Subjects must agree to not use high-dose aspirin during the course of the study. Daily low-dose aspirin treatment (not more than 81 mg per day) may be continued if currently prescribed.
9. requiring long-term glucocorticoid therapy or chronic immunosuppressive therapy; Inhaled steroid use for management of asthma is not an absolute exclusion.
10. use of lithium
11. participation in an experimental medication trial within 3 months of starting the study;
12. current therapy for malignant disease other than basal- cell or squamous-cell skin cancer;
13. history of gastrointestinal bleeding or active gastric ulcer; screening laboratory abnormalities including AST (SGOT) and or ALT (SGPT) > 2.5 x the upper limit of normal (ULN), total bilirubin > 1.5 x ULN, platelets < 100,000;
14. You have developed keloid scarring in the past. Keloids are large, thick masses of scar tissue. These are more common among dark-skinned people.
15. presence of any condition that, in the opinion of the investigator would make it unlikely for the subject to complete 12 months of study participation, e.g., history of non- adherence to therapeutic regimens, presence of conditions likely to limit life expectancy, living situation that would interfere with study visit schedules such as a job requiring frequent or extended travel
16. known hypersensitivity to salsalate. Patients who have experienced asthma, hives, or other allergic-type reactions to aspirin or other NSAIDs are excluded from participation. Patients with known or suspected aspirin or NSAID-sensitive asthma are excluded.

In addition, subjects with concurrent chicken pox, influenza, flu-like symptoms or other symptomatic viral illnesses should not be enrolled in the study until the illness or condition has resolved.

Subjects with known or suspected hypersensitivity to lidocaine or epinephrine may not be able to participate as these agents are used for local anesthesia during skin biopsies. The study investigators should consider the nature and severity of past reported reactions to these agents, and may consider alternative anesthesia options for local anesthesia on a case by case basis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-10; Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Pop-Busui, MD, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Veterans Administration Ann Arbor Health Center, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ang L, Gunaratnam S, Huang Y, Dillon BR, Martin CL, Burant A, Reiss J, Blakely P, Vasbinder A, Zhao L, Mizokami-Stout K, Tang Y, Feldman EL, Doria A, Spino C, Banerjee M, Hayek SS, Pop-Busui R. Inflammatory Markers and Measures of Cardiovascular Autonomic Neuropathy in Type 1 Diabetes. J Am Heart Assoc. 2025 Jan 7;14(1):e036787. doi: 10.1161/JAHA.124.036787. Epub 2024 Dec 27. PMID 39727210

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ninety-six (96) people underwent eligibility screening to participate in the study. Of these, 64 satisfied the eligibility criteria for participation, and 61 were randomly assigned and entered the treatment phase of the study (and shown as started in the table below). Three of the 64 eligible participants did not complete visit 2, and therefore, were not assigned to treatment. Informed consent was obtained from all participants at the time of their screening visit.
Period: Overall Study
Arm/Group | Salsalate | Comparator
Started | 37 | 24
Completed | 33 | 22
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Salsalate | Comparator | Total
Number analyzed (Participants) | 37 | 24 | 61
Age, Continuous [Mean (Full Range); unit: years] | 48.8 [21 to 70] | 51.9 [34 to 69] | 51.5 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 21 | 13 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 33 | 24 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 36 | 23 | 59
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 24 | 61

OUTCOME MEASURES:

1. Primary Outcome: Skin Biopsy - Intraepidermal Nerve Fiber Density (IENFD) - Distal Thigh
Description: The intraepidermal nerve fiber density (IENFD) is the number of small nerve fibers which can be counted (under a microscope) in a 3 mm piece of skin taken from the distal (lower) thigh. IENFD is a continuous measure of small fiber neuropathy, with high positive and negative predictive values along with a high diagnostic efficiency in differentiating between people with and without neuropathy. People with neuropathy will generally have fewer nerve fibers (lower IENFD) than people without neuropathy. This study examined the change in IENFD after taking salsalate or a placebo daily for 12 months in people with diabetic neuropathy. Skin samples taken at the start of the study were compared to skin samples taken 12 months later to see if salsalate caused an increase in IENFD (suggesting improvement), or smaller decrease in IENFD (suggesting slower progression of neuropathy) relative to placebo.
Time Frame: 12 months
Population: The analysis is limited to participants with analyzable skin samples at both baseline and at 12 months. Participants who withdrew or were lost to follow-up prior to 12 months are not included in this analysis.
Measure: Mean (Standard Deviation); unit: Percentage change in IENFD
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 33 | 22
Percentage change in IENFD | 12 (57) | 14 (55)

2. Secondary Outcome: Measures of Cardiac Autonomic Neuropathy (CAN) - Valsalva Ratio
Description: Valsalva Ratio is the ratio of max tachycardia to max bradycardia caused by Valsalva maneuver
Time Frame: Baseline and 12 Months
Population: This analysis is limited to participants who completed the valsalva maneuver successfully at both the baseline and final study visits. Participants who withdrew (N=2) or were lost to follow-up (4) are not included in the analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 33 | 22
ratio
  Baseline - Valsalva Ratio | 2.81 (1.18) | 2.29 (0.66)
  12 Month - Valsalva Ratio | 2.73 (1.12) | 2.37 (0.93)

3. Secondary Outcome: Measures of Cardiac Autonomic Neuropathy (CAN) - Expiration/Inspiration Ratio
Description: The expiration/inspiration ratio (E/I) ratio is measured during a period of slow, deep breathing (6 breaths per minute). It is the average heart rate increase divided by the average heart rate decrease over 6 breath cycles per minute
Time Frame: Baseline and 12 Months
Population: Only participants with both baseline and 12 month data were included in analysis. Participants who withdrew (N=2) or were lost to follow-up (N=4) are not included in the analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 33 | 22
ratio
  Baseline - E/I Ratio | 1.14 (0.12) | 1.12 (0.1)
  12 Months - E/I Ratio | 1.21 (0.5) | 1.11 (0.08)
Statistical Analysis 1: Comparison: Salsalate vs Comparator; TTEST, two sided; Test type: Superiority; p = 0.41, t-test, 2 sided; 2-sided

4. Secondary Outcome: Measures of Cardiac Autonomic Neuropathy (CAN) - 30:15 Ratio
Description: Ratio of max RR interval ~30 heartbeats to min RR interval ~15 heartbeats
Time Frame: Baseline and 12 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 33 | 22
ratio
  Baseline - 30:15 Ratio | 1.15 (0.1) | 1.12 (0.1)
  12 Month - 30:15 Ratio | 1.39 (1.55) | 1.10 (0.08)

5. Secondary Outcome: Measures of Cardiac Autonomic Neuropathy (CAN) - SDNN
Description: Standard deviation of NN intervals. The value indicates the amount of variability in the interval between each heart beat (the R-R interval). Value is expressed in milliseconds
Time Frame: Baseline and 12 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 33 | 22
milliseconds
  Baseline - SDNN | 39 (23) | 36 (31)
  12 Month - SDNN | 47 (49) | 35 (26)

6. Secondary Outcome: Measures of Cardiac Autonomic Neuropathy (CAN) - RMSSD
Description: Root mean square of successive differences between normal heartbeats. It represents the average variation between the beat to beat intervals. The result is expressed in milliseconds.
Time Frame: Baseline and 12 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 33 | 22
milliseconds
  Baseline - RMSSD | 24 (16) | 22 (22)
  12 Month - RMSSD | 33 (47) | 20 (20)

7. Secondary Outcome: Nerve Conduction
Description: Nerve Conduction Studies of the sural, peroneal, and ulnar nerves will be obtained at screening and 12 months. Nerve conduction studies are used to detect abnormalities in how the nerves are working. Nerve Conduction is represented as number of nerves with abnormal nerve conduction per participant.
Time Frame: Baseline and 12 months
Population: All participants are included in the baseline analysis. Data are not available for participants who withdrew (N=2) or were lost to follow-up (4) prior to month 12, and for one additional participant who was unwilling to undergo the nerve conduction test at the final study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 37 | 24
Participants
  Baseline: Participants with 0 Abnormal Nerves | 1 | 1
  Baseline: Participants with 1 Abnormal Nerve | 9 | 2
  Baseline: Participants with 2 Abnormal Nerves | 5 | 2
  Baseline: Participants with 3 Abnormal Nerves | 22 | 19
  12 months: number analyzed (Participants) | 32 | 22
  12 months: Participants with 0 Abnormal Nerves | 1 | 3
  12 months: Participants with 1 Abnormal Nerve | 5 | 1
  12 months: Participants with 2 Abnormal Nerves | 10 | 1
  12 months: Participants with 3 Abnormal Nerves | 16 | 17

8. Secondary Outcome: Quantitative Sensory Testing - Just Noticeable Difference in COLD Detection
Description: The Just Noticeable Difference (JND) in response to a cold stimulus applied to the top of the foot was measured using the CASE IV System. The range of JND values is from 1 to 25. A JND value of 1 means a person can detect temperature decrease of 0.063 degrees Celsius while a JND value of 25 means that the temperature has to drop by 20 degrees Celsius colder than before the person can notice the change in temperature. People with neuropathy will have higher JND values than people without neuropathy, indicating that they are less able to detect changes in temperature. For this study, the cold JND at the first visit was compared to the JND at the second visit to see if JND for cold detection after 12 months of treatment with salsalate or placebo.
Time Frame: Baseline and 12 months
Population: Two enrolled participants are missing baseline data for this specific outcome measure as the device (CASE IV) could not record a response (technical limitations). The 12 month data excludes participants who withdrew (N=2) or were lost to follow up (N=4), one participant who declined the test at study end, and excludes results for 5 participants due to technical limitations of the device.
Measure: Mean (Standard Deviation); unit: JND Units
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 36 | 23
JND Units
  Baseline | 14.67 (5.12) | 16.46 (4.25)
  12 Month: number analyzed (Participants) | 31 | 18
  12 Month | 13.56 (5.53) | 14.37 (5.11)

9. Secondary Outcome: Quantitative Sensory Testing - Just Noticeable Difference- Vibration
Description: The Just Noticeable Difference (JND) in response to a vibrating stimulus (probe) applied to the toe was measured using the CASE IV System. The range of JND values is from 1 to 25. A JND value of 1 means a person can detect very light vibration (vibration magnitude of 0.106 micrometers) while a 25 means a much stronger vibration stimulus had to be applied to be detected (vibration magnitude of 576.603 micrometers). People with neuropathy will have higher JND values than people without neuropathy, indicating that they are less able to detect vibration. For this study, the vibration JND at the first visit was compared to the vibration JND at the second visit to see if the values had changed after 12 months.
Time Frame: Baseline and 12 months
Population: Three enrolled participants (of 61 total enrolled) are missing baseline data for this specific measure as the CASEIV device could not record a response (technical limitations). The 12 month data excludes participants who withdrew (N=2) or were lost to follow up (N=4), one participant who declined the test at study end, and for 4 participants due to technical limitations of the CASE IV device.
Measure: Mean (Standard Deviation); unit: JND Units
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 36 | 22
JND Units
  Baseline | 18.91 (3.0) | 19.62 (3.26)
  12 Month: number analyzed (Participants) | 31 | 19
  12 Month | 19.62 (3.46) | 20.38 (2.55)

10. Secondary Outcome: Diabetic Neuropathy Symptoms
Description: DN symptoms as evaluated by the Neuropathy Total Symptom Score-6 (NTSS-6). The NTSS-6 has 6 questions with individual scores between 0 and 3.66. Cumulative scores range from 0 to 21.96 with 21.96 being the worst neuropathy and 0 being no neuropathy.
Time Frame: Baseline to 12 months
Population: Baseline data is available for all enrolled participants. 12 months data excludes participants who withdrew (N=2),or were lost to follow-up (N=4) and 2 participants with incomplete or missing surveys at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 37 | 24
score on a scale
  Baseline | 4.5 (4.2) | 4.6 (3.1)
  12 Month: number analyzed (Participants) | 32 | 21
  12 Month | 3.3 (4.1) | 4.2 (4.2)

11. Secondary Outcome: Survey of Autonomic Symptoms (SAS)
Description: Survey of Autonomic Symptoms (SAS) is a 12-item questionnaire. The range of scores is 0-60 for men and 0-55 for women, with higher scores indicating a higher degree of autonomic symptoms. Men and Women were not analyzed separately due to the comparable gender distribution between arms.
Time Frame: Baseline to 12 months
Population: Baseline data is available for all enrolled participants. 12 months data excludes participants who withdrew (N=2), or were lost to follow-up (N=4) and 2 participants with incomplete or missing surveys at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 37 | 24
score on a scale
  Baseline | 3.6 (2.2) | 3.9 (1.8)
  12 Months: number analyzed (Participants) | 32 | 21
  12 Months | 3.4 (2.3) | 2.9 (2.0)

12. Secondary Outcome: The DCCT/EDIC Structured Neurological Examination
Description: The DCCT/EDIC Structured Neurological Examination is an examination that determines whether or not someone has evidence of neuropathy from diabetes. The examination categorizes patients into 3 categories: Definite Clinically Evident Peripheral Neuropathy, Possible Clinically Evident Peripheral Neuropathy, and No Clinically Evident Peripheral Neuropathy.
Time Frame: Baseline and 12 months
Population: Baseline data is available for all enrolled participants. 12 months data excludes participants who withdrew (N=2), or were lost to follow-up (N=4) and 2 participants who did not complete the examination at the 12 month time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 37 | 24
Participants
  Baseline: Definite Clinically Evident Peripheral Neuropathy | 27 | 20
  Baseline: Possible Clinically Evident Peripheral Neuropathy | 10 | 3
  Baseline: No Clinically Evident Peripheral Neuropathy | 0 | 1
  12 Months: number analyzed (Participants) | 32 | 21
  12 Months: Definite Clinically Evident Peripheral Neuropathy | 28 | 21
  12 Months: Possible Clinically Evident Peripheral Neuropathy | 4 | 0
  12 Months: No Clinically Evident Peripheral Neuropathy | 0 | 0

13. Secondary Outcome: NeuroQOL
Description: NeuroQOL is a self-administered questionnaire that measures the impact of neuropathy symptoms, especially those affecting the feet and legs, on quality of life. Shown are results from baseline, 6 and 12 months for the item "Overall, I would say problem with my feet reduced my quality of life". Responses are on a five-point scale (1 = "not at all" up to 5 = "very much") with higher values indicating a greater reduction in quality of life.
Time Frame: Baseline, 6 months and 12 months
Population: The survey was completed by all enrolled participants at baseline. Six (6) and 12 month values are shown for all participants who had not withdrawn from the study or were lost to follow-up prior to the survey administration. One participant who completed the study, did not complete the survey at month 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 37 | 24
score on a scale
  Baseline | 1.9 (1.1) | 1.8 (1.0)
  6 Months: number analyzed (Participants) | 35 | 22
  6 Months | 1.74 (0.98) | 1.77 (0.92)
  12 Months: number analyzed (Participants) | 32 | 21
  12 Months | 1.8 (1.0) | 2.1 (1.2)

14. Secondary Outcome: Neuropathic Pain Scale
Description: The Neuropathic Pain Scale is a questionnaire where participants rate the intensity of their pain and the quality of the pain (e.g., burning, aching, stabbing). Higher scores indicate greater pain. Scores range from 0 to 100.
Time Frame: baseline, 6 months, 12 months
Population: Baseline data is available for all enrolled participants. Six (6) and12 month data excludes those participants who had withdrawn, or had been declared lost to follow-up prior to the visit at which the survey was administered.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 37 | 24
score on a scale
  Baseline | 30.95 (20.98) | 29.21 (20.29)
  6 Month: number analyzed (Participants) | 35 | 22
  6 Month | 27.06 (19.89) | 28.36 (20.31)
  12 Month: number analyzed (Participants) | 33 | 21
  12 Month | 27.06 (20.70) | 28.86 (18.72)

15. Secondary Outcome: The Berg Balance Scale
Description: The Berg Balance Scale measures balance in 14 separate activities of daily living such as going from sitting-to-stand and standing on one leg; the unipedal stance portion that had been shown to be particularly reflective of neuropathy-related mobility loss. Scores range from 0 to 56, where lower scores indicate worst mobility and balance and 56 indicates best mobility and balance.
Time Frame: Baseline and 12 months
Population: Data from all enrolled participants is shown at baseline. The 12 month data excludes patients who had withdrawn (N=2) or were lost to follow-up (N=4), and an additional two participants who did not complete measure at the final visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 37 | 24
score on a scale
  Baseline | 54.6 (2.6) | 53.8 (2.3)
  12 Months: number analyzed (Participants) | 32 | 21
  12 Months | 55.3 (1.3) | 52.7 (8.2)

16. Secondary Outcome: 8 Foot Up and Go Test
Description: The 8 Foot Up and Go Test, a test of functional mobility that assesses the time needed for a subject to arise from sitting position, walk 8 ft and turn 180 degrees around a cone and return sitting; Test results are expressed in seconds. The test is performed twice and the fastest speed is reported.
Time Frame: Baseline and 12 months
Population: Baseline analysis includes all enrolled participants. The final visit analysis excludes participants who withdrew (N = 2) or were lost to follow-up (N=4), and 2 participants who did not complete the measure at their final study visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 37 | 24
seconds
  Baseline | 5.60 (1.63) | 5.78 (1.17)
  12 Month: number analyzed (Participants) | 33 | 20
  12 Month | 5.56 (1.07) | 5.90 (1.26)

17. Secondary Outcome: The Modified Falls Efficacy Scale
Description: The Modified Falls Efficacy Scale assessing patient's self-reported ability to perform activities of daily living (e.g. get dressed/ undressed, walking, shopping). Scores range from 0 to 10 on 14 items. Resulting score is average score across those 14 questions, resulting in a score from 0 to 10. 0 represents the participant being not at all confident that they can complete activities without falling and 10 represents participant being entirely confident that they can complete activities without falling.
Time Frame: Baseline and 12 months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Salsalate | Comparator
Number analyzed (Participants) | 37 | 24
score on a scale
  Baseline | 9.4 (1.3) | 9.2 (1.3)
  12 Months: number analyzed (Participants) | 32 | 21
  12 Months | 9.5 (1.2) | 9.1 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at each participant visit starting from screening (Visit 1) to the final study visit (Visit 7), typically about 12 months.
Description: Adverse event reporting is described in the protocol.
Arm/Group | Salsalate | Comparator
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/24
Serious Adverse Events (participants affected / at risk) | 6/37 | 4/24
Other Adverse Events (participants affected / at risk) | 30/37 | 19/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salsalate (N=37) | Comparator (N=24)
CARDIOVASCULAR EVENTS (Cardiac disorders) | 3 (3) | 1 (1)
HYPERGLYCEMIA/DIABETIC KETOACIDOSIS (Endocrine disorders) | 2 (3) | 1 (1)
NAUSEA AND VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) — SEVERE NAUSEA AND VOMITING IN PATIENT WITH KNOWN GASTROPARESIS
ALLERGIC REACTION (Immune system disorders) | 0 (0) | 1 (1) — SEVERE ALLERGIC REACTION TO LAUNDRY SOAP
INFECTION (Infections and infestations) | 2 (3) | 0 (0)
INJURY (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Salsalate (N=37) | Comparator (N=24)
Endocrine, Endocrine/Infectious, Endocrine/Gastrointestinal (Endocrine disorders) | 5 | 7
Cardiac, Cardiovascular, Circulatory disorders (Cardiac disorders) | 4 | 1
Gastrointestinal adverse event (Gastrointestinal disorders) | 12 | 4
Infection (Infections and infestations) | 15 | 4
Musculoskeletal adverse event (Musculoskeletal and connective tissue disorders) | 7 | 7
Otorhinolaryngologic adverse event (Ear and labyrinth disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT02936843/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT02936843/ICF_000.pdf